CLINICAL TRIAL: NCT05509452
Title: Risk Factors of Incisional Hernias After Emergency Midline Laparotomy: a Danish Prospective Single-center, Non-randomized, Non-interventional, Descriptive Follow-up Study
Brief Title: Risk Factors of Incisional Hernias After Emergency Midline Laparotomy
Acronym: INCISE
Status: Not yet recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Madeline Kvist, Principal Investigator, Herlev Hospital
Other Study IDs: HerlevH1
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Incisional Hernia; Emergency Midline Laparotomy
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify risk factors for the development of incisional hernias in emergency midline laparotomies.

DETAILED DESCRIPTION:
All patients operated with an emergency midline laparotomy and attending 1-year follow-up in our clinic is potential participants and will be screened for participation. Potential participants will be briefly informed about the project by the hospital staff. If the patients are interested, they will be thoroughly informed about the study and asked to participate by one of the trial investigators before discharge.

Data will be obtained from the participants hospital files and by patient survey/interview. All data will be entered into a database using RedCap by trial investigators or their delegates.

Enrolled patients will be followed for two years. The trial involves two clinical examinations and evaluations (one and two years) after surgery. Clinical examination involves interview with a standardized questionnaire and abdominal wall examination including inspection, palpation and ultrasound examination.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or above and
* Unscheduled midline laparotomy in an emergency or subacute setting, involving perforated bowel, bowel obstruction, bowel ischemia (due to mesenteric vascular disease or incarceration), inflammatory diseases (e.g. diverticulitis, appendicitis, ulcerative colitis, cholecystitis and Crohn's disease), abscesses, non-traumatic intraabdominal bleeding and any emergency re-operation to elective surgery

Exclusion Criteria:

* Age below 18 years
* Patients with mental or physical disorders making follow-up impossible
* Patients were no fascial closure is performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient operated with an emergency midline laparotomy and followed up in our clinic will be evaluated for enrollment. Patients will be eligible if they comply with the inclusion and exclusion criteria listed above.
  We aim to include a total of 500 patients for the first follow-up. This is based on a drop out and long-term death of approximately 50%, incisional hernia rate of 20% and 10 risk factors in multivariate analysis requiring 100 patients with incisional hernias. 100 incisional hernias = 500 patients included at first post-operative follow up.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Risk factors of incisional hernia after emergency midline laparotomy | 2 years
  Multivariate analysis on selected variables evaluated for long-term complications, including sex, age, high BMI, active smoking, hernia in the midline, length of incision, rectus muscle diastasis, sarcopenia, peritonitis and multiple laparotomies

SECONDARY OUTCOMES:
Rate of incisional hernias one and two years after surgery | 2 years
30-day, 90-day, 1-year and 2-year mortality | 2 years
Rates of asymptomatic versus symptomatic incisional hernias | 2 years
Rate of surgery for incisional hernias 2-years post index surgery | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal- and Hepatic diseases, Surgical Section,, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All results, both positive, negative and inconclusive, will be attempted to be published in international English journals with external reviewers. Alternatively, the results will be published in another way.
Supporting Information: Study Protocol, ICF, CSR